CLINICAL TRIAL: NCT02983500
Title: Tablet-based Prospective Patient Reported Outcomes (PRO) Registry in Patients With Advanced NSCLC or Advanced Pancreatic Cancer With Focus on Cancer Cachexia
Brief Title: Patient Reported Outcomes Registry in Patient With Cancer Cachexia
Acronym: PROXie
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Chugai Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-0050346
Record Dates: First submitted 2016-10-24; First posted 2016-12-06 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Metastatic Pancreatic Cancer; NSCLC, Metastatic
Keywords: Patient Reported Outcome (PRO)
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluation of patient reported outcomes (PRO) with tumor cachexia in a real life setting.

DETAILED DESCRIPTION:
The PRO Xie project will recruit a representative cohort of patients with advanced lung or advanced pancreatic cancer with a high risk for the development of cancer cachexia.

Patient Reported Outcomes (PRO) are assessed in a real life setting by a questionnaire consisting of 20 questions: QoL is measured by SF12, fatigue by FACIT-F and cachexia by FAACT questionnaires, respectively.

These data will determine the potential need for anti-cachexia treatment in those patients, as well as the number of underweight patients, the evaluation of general QoL, fatigue and cachexia and the evaluation of malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of NSCLC UICC stage IIIB/IV or pancreatic cancer UICC stage III/IV
* Start of the first line palliative systemic treatment
* Ability to read and understand German
* Written informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with locally advanced and unresectable or metastatic NSCLC (UICC Stage IIIB/IV) or locally advanced and unresectable or metastatic pancreatic cancer (UICC stage III/IV) at start of their first-line palliative systemic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2016-08-28 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Rate of patients with loss of > 5 % body weight | 18 months

SECONDARY OUTCOMES:
Number of underweight patients | 12 months
  BMI < 20 kg/qm at start or during observation.
General health-related quality of life assessment | 12 months
  At baseline, throughout and at the end of the study with SF 12 questionnaire.
Fatigue assessment | 12 months
  At baseline, throughout and at the end of the study with FACIT-F (short version of fatigue subscale).
Cachexia assessment | 12 months
  At baseline, throughout and at the end of the study with FAACT (short version of anorexia / cachexia subscale).

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Welslau, MD, Principal Investigator — Medical practise for oncology
Locations (1):
- Multiple sites all over Germany, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: No